CLINICAL TRIAL: NCT02343120
Title: A Phase I/II, Open-Label, Multiple-Dose, Dose Escalation and Expansion Study to Investigate the Safety and Pharmacokinetics of the BTK Inhibitor BGB-3111 in Subjects With B-Cell Lymphoid Malignancies
Brief Title: Study of the Safety and Pharmacokinetics of BGB-3111 in Subjects With B-Cell Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-AU-003; 2016-003364-39 (EudraCT Number)
Record Dates: First submitted 2015-01-09; First posted 2015-01-21 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: B-cell Malignancies
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Participants were administered up to 320 mg total daily dose of zanubrutinib until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Oral administration by capsule
  Other Names: BGB-3111; Brukinsa

SUMMARY:
This study evaluated the safety, tolerability, pharmacokinetic profile and efficacy of BGB-3111 in participants with B-cell lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years, voluntarily consented to the study.
2. WHO classification defined B-lymphoid malignancy, with the exception of Burkitt lymphoma/leukemia, plasma cell myeloma, acute lymphoblastic leukemia, lymphoblastic lymphoma, and plasmablastic lymphoma.
3. Requirement for treatment in the opinion of the investigator.
4. Disease which has relapsed, or is refractory, following at least one line of therapy, with no therapy of higher priority available.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Adequate hematologic function, as defined by neutrophils ≥ 1.0 x 10^9/L and platelets ≥ 50 x 10^9/L; participants with neutrophils < 1.0 x 10^9/L due to marrow infiltration are allowed to receive growth factors to bring pre-treatment neutrophils to ≥ 1.0 x 10^9/L.
7. Adequate renal function, as defined by creatinine clearance of ≥ 30 ml/min (as estimated by the Cockcroft-Gault equation or as measured by nuclear medicine scan or 24 hour urine collection).
8. Adequate liver function, as defined by aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN), and bilirubin ≤ 1.5 x ULN (unless documented Gilbert's syndrome).
9. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN.
10. Female participants of childbearing potential and non-sterile males must practice at least one of the following methods of birth control with partner(s) throughout the study and for 90 days after discontinuing study drug: total abstinence from sexual intercourse, double-barrier contraception, IUD or hormonal contraceptive initiated at least 3 months prior to first dose of study drug.
11. Male participants must not donate sperm from initial study drug administration, until 90 days after drug discontinuation.

Exclusion Criteria:

1. Current central nervous system (CNS) involvement by disease
2. Current histologically transformed disease.
3. Prior Bruton's tyrosine kinase (BTK) inhibitor treatment.
4. Allogeneic stem cell transplantation within 6 months, or has active graft-versus-host disease (GVHD) requiring ongoing immunosuppression.
5. Receipt of the following treatment prior to first dose of zanubrutinib: corticosteroids given with anti-neoplastic intent within 7 days, chemotherapy or radiotherapy within 2 weeks, monoclonal antibody within 4 weeks.
6. Not recovered from toxicity of any prior chemotherapy to grade ≤ 1.
7. History of other active malignancies within 2 years of study entry, with exception of (1) adequately treated in-situ carcinoma of cervix; (2) localized basal cell or squamous cell carcinoma of skin; (3) previous malignancy confined and treated locally (surgery or other modality) with curative intent.
8. Uncontrolled systemic infection requiring parenteral anti-microbial therapy.
9. Major surgery in the past 4 weeks.
10. Known HIV, or active hepatitis B or hepatitis C infection (detected positive by PCR).
11. Cardiovascular disease resulting in New York Heart Association function status of ≥ 3.
12. Significant active renal, neurologic, psychiatric, hepatic or endocrinologic disease that in the investigator's opinion would adversely impact on his/her participating in the study.
13. Inability to comply with study procedures.
14. On medications which are cytochrome P450 (CYP) 3A inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (23):
- United States (4):
  - Banner MD Anderson Cancer Centre, Gilbert, Arizona
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - M.D. Anderson Cancer Center, Houston, Texas
- Australia (11):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Parkville, Victoria
  - Melbourne Health, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Italy (2):
  - Policlinico S.Orsola Malpighi, AOU di Bologna, Bologna
  - Ospedale Maggiore Policlinico, Fondazione IRCCS Ca' Granda, Milan
- North Shore Hospital, Auckland, New Zealand
- South Korea (4):
  - Dong-A University Medical Centre, Busan
  - Inje University Busan Paik Hospital, Busan
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
- Derriford Hospital, Plymouth, Devon, United Kingdom

REFERENCES:
- [Background] Tam CS, Trotman J, Opat S, Burger JA, Cull G, Gottlieb D, Harrup R, Johnston PB, Marlton P, Munoz J, Seymour JF, Simpson D, Tedeschi A, Elstrom R, Yu Y, Tang Z, Han L, Huang J, Novotny W, Wang L, Roberts AW. Phase 1 study of the selective BTK inhibitor zanubrutinib in B-cell malignancies and safety and efficacy evaluation in CLL. Blood. 2019 Sep 12;134(11):851-859. doi: 10.1182/blood.2019001160. Epub 2019 Jul 24. PMID 31340982
- [Background] Trotman J, Opat S, Gottlieb D, Simpson D, Marlton P, Cull G, Munoz J, Tedeschi A, Roberts AW, Seymour JF, Atwal SK, Yu Y, Novotny W, Holmgren E, Tan Z, Hilger JD, Huang J, Tam CS. Zanubrutinib for the treatment of patients with Waldenstrom macroglobulinemia: 3 years of follow-up. Blood. 2020 Oct 29;136(18):2027-2037. doi: 10.1182/blood.2020006449. PMID 32698195
- [Background] C.S. Tam M. Wang D. Simpson S. Opat G. Cull J. Munoz T.J. Phillips W. Kim S. Atwal R. Wei J. Huang R. Elstrom J. Trotman. UPDATED SAFETY AND EFFICACY DATA IN THE PHASE 1 TRIAL OF PATIENTS WITH MANTLE CELL LYMPHOMA (MCL) TREATED WITH BRUTON TYROSINE KINASE (BTK) INHIBITOR ZANUBRUTINIB (BGB-3111). Hematological Oncology. 2019; 37(S2) DOI: https://doi.org/10.1002/hon.55_2630
- [Background] Cull G, Burger JA, Opat S, Gottlieb D, Verner E, Trotman J, Marlton P, Munoz J, Johnston P, Simpson D, Stern JC, Prathikanti R, Wu K, Novotny W, Huang J, Tam CS. Zanubrutinib for treatment-naive and relapsed/refractory chronic lymphocytic leukaemia: long-term follow-up of the phase I/II AU-003 study. Br J Haematol. 2022 Mar;196(5):1209-1218. doi: 10.1111/bjh.17994. Epub 2021 Dec 16. PMID 34915592
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Xu W, Yang S, Tam CS, Seymour JF, Zhou K, Opat S, Qiu L, Sun M, Wang T, Trotman J, Pan L, Gao S, Zhou J, Zhou D, Zhu J, Song Y, Hu J, Feng R, Huang H, Su D, Shi M, Li J. Zanubrutinib Monotherapy for Naive and Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma: A Pooled Analysis of Three Studies. Adv Ther. 2022 Sep;39(9):4250-4265. doi: 10.1007/s12325-022-02238-7. Epub 2022 Jul 28. PMID 35900694
- [Derived] Phillips T, Chan H, Tam CS, Tedeschi A, Johnston P, Oh SY, Opat S, Eom HS, Allewelt H, Stern JC, Tan Z, Novotny W, Huang J, Trotman J. Zanubrutinib monotherapy in relapsed/refractory indolent non-Hodgkin lymphoma. Blood Adv. 2022 Jun 14;6(11):3472-3479. doi: 10.1182/bloodadvances.2021006083. PMID 35390135
- [Derived] Tam CS, Opat S, Simpson D, Cull G, Munoz J, Phillips TJ, Kim WS, Rule S, Atwal SK, Wei R, Novotny W, Huang J, Wang M, Trotman J. Zanubrutinib for the treatment of relapsed or refractory mantle cell lymphoma. Blood Adv. 2021 Jun 22;5(12):2577-2585. doi: 10.1182/bloodadvances.2020004074. PMID 34152395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts. The dose escalation part (Part 1) determined the recommended phase 2 dose (RP2D) and regimen and the dose expansion part (Part 2) further characterized the safety and efficacy at the RP2D.
Groups:
- Part 1: 40 mg QD: Participants received 40 mg of zanubrutinib once daily (QD) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up
- Part 1: 80 mg QD: Participants received 80 mg of zanubrutinib once daily (QD) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up
- Part 1: 160 mg QD: Participants received 160 mg of zanubrutinib once daily (QD) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up
- Part 1 and Part 2: 160 mg BID: Part 1: Participants received 160 mg of zanubrutinib twice daily (BID) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up were evaluated. Part 2: This dose regimen was selected for further evaluation in various expansion cohorts that span multiple disease types.
- Part 1 and Part 2: 320 mg QD: Part 1: Participants received 320 mg of zanubrutinib once daily (QD) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up were evaluated. Part 2: This dose regimen was selected for further evaluation in various expansion cohorts that span multiple disease types.
Period: Part 1: Dose Escalation
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Started | 3 | 4 | 5 | 4 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 5 | 4 | 1
Not completed — Sponsor decision | 1 | 2 | 3 | 2 | 0
Not completed — Death | 1 | 2 | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Period: Part 2: Expansion
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Started | 0 | 0 | 0 | 274 | 94
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 274 | 94
Not completed — Sponsor decision | 0 | 0 | 0 | 165 | 67
Not completed — Death | 0 | 0 | 0 | 74 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 28 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5 | 2
Not completed — Other | 0 | 0 | 0 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD | Total
Number analyzed (Participants) | 3 | 4 | 5 | 278 | 95 | 385
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (9.45) | 62.3 (14.38) | 72.6 (8.88) | 66.4 (11.21) | 65.8 (11.24) | 66.3 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 86 | 20 | 109
  Male | 2 | 3 | 4 | 192 | 75 | 276
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 2 | 4 | 5 | 205 | 87 | 303
  Asian | 1 | 0 | 0 | 47 | 5 | 53
  Black or African American | 0 | 0 | 0 | 4 | 1 | 5
  Native Hawaiians or other Pacific Islanders | 0 | 0 | 0 | 2 | 0 | 2
  Multiple | 0 | 0 | 0 | 1 | 0 | 1
  Not Reported | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 18 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and Part 2: Number of Participants With Adverse Events
Description: Number of participants with adverse events and serious adverse events, including clinically relevant physical examinations and laboratory measurements
Time Frame: Up to approximately 6 years and 7 months
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Parts 1 and 2: 160 mg BID: Part 1: Participants received 160 mg of zanubrutinib twice daily (BID) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up. Part 2: This dose regimen was selected for further evaluation in various expansion cohorts that span multiple disease types.
- Parts 1 and 2: 320 mg QD: Part 1: Participants received 320 mg of zanubrutinib once daily (QD) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up. Part 2: This dose regimen was selected for further evaluation in various expansion cohorts that span multiple disease types.
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Parts 1 and 2: 160 mg BID | Parts 1 and 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 278 | 95
Participants
  At least one treatment-emergent adverse event | 3 | 4 | 5 | 274 | 94
  Serious adverse events | 1 | 2 | 3 | 157 | 45

2. Primary Outcome: Part 1: Recommended Phase 2 Dose (RP2D) for Zanubrutinib
Description: RP2D for zanubrutinib was the maximum tolerated dose (MTD) or less, which was determined by testing increasing doses up to 320 mg QD
Time Frame: Month 9
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of study drug
Measure: Number; unit: milligrams
Groups:
- Part 1: Zanubrutinib: Five dose regimens of zanubrutinib (40 mg QD, 80 mg QD, 160 mg QD, 160 mg BID, and 320 mg QD) were evaluated.
Arm/Group | Part 1: Zanubrutinib
Number analyzed (Participants) | 17
milligrams | 320

3. Secondary Outcome: Part 1 and Part 2: Area Under the Curve From Time 0 to the Last Sampling Time Point Within the Dose Interval (AUClast) of Zanubrutinib
Time Frame: Week 1 Day 1 pre-dose, 0.5, 1, 2, 3, 4, and 8 hours
Population: The pharmacokinetic (PK) analysis set included all participants for whom valid zanubrutinib PK parameters could be estimated, shown as overall number analyzed. Only participants with available data per dose were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters*hour
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Parts 1 and 2: 160 mg BID | Parts 1 and 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 76 | 19
nanograms/milliliters*hour | 274.7 (47.8) | 436.8 (103.5) | 1480 (53.0) | 1132 (61.1) | 2281 (60.5)

4. Secondary Outcome: Part 1 and Part 2: Area Under the Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Zanubrutinib
Time Frame: Week 1 Day 1 pre-dose, 0.5, 1, 2, 3, 4, and 8 hours
Population: The PK analysis set included all participants for whom valid zanubrutinib PK parameters could be estimated, shown as overall number analyzed. Only participants with available data per dose were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters*hour
Groups:
- Part 1 and Part 2: 160 mg BID: Part 1: Participants received 160 mg of zanubrutinib twice daily (BID) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up. Part 2: This dose regimen was selected for further evaluation in various expansion cohorts that span multiple disease types.
- Part 1 and Part 2: 320 mg QD: Part 1: Participants received 320 mg of zanubrutinib once daily (QD) orally until disease progression, intolerance or death, withdrawal of consent, or loss to follow-up. Part 2: This dose regimen was selected for further evaluation in various expansion cohorts that span multiple disease types.
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 59 | 18
nanograms/milliliters*hour | 301.1 (51.5) | 460.0 (100.6) | 1505 (52.7) | 1253 (59.0) | 2538 (47.8)

5. Secondary Outcome: Part 1 and Part 2: Maximum Observed Plasma Concentration (Cmax) After Administration of Zanubrutinib
Time Frame: Week 1 Day 1 pre-dose, 0.5, 1, 2, 3, 4, and 8 hours
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Groups:
- Part 1: 160 mg QD: Participants received 160 mg of zanubrutinib once daily (QD) orally until disease progression, intolerance or death, withdrawal of consent, or loss to
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 76 | 19
nanograms/milliliter | 86.0 (46.6) | 125 (77.6) | 397 (76.1) | 304 (63.8) | 566 (65.6)

6. Secondary Outcome: Part 1 and Part 2: Maximum Observed Plasma Concentration (Cmax) After Administration of Zanubrutinib
Time Frame: Week 2 Day 1 pre-dose and 24 hours
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 77 | 72
nanograms/milliliter | 75.7 (36.2) | 169 (50.0) | 387 (60.7) | 299 (56.1) | 533 (55.0)

7. Secondary Outcome: Part 1 and Part 2: Time to Maximum Observed Plasma Concentration (Tmax) of Zanubrutinib
Time Frame: Week 1 Day 1 pre-dose, 0.5, 1, 2, 3, 4, and 8 hours
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 76 | 19
Hours | 1.00 [0.50 to 1.98] | 2.00 [1.17 to 2.00] | 1.92 [0.93 to 2.08] | 2.00 [0.83 to 8.00] | 2.00 [0.72 to 3.08]

8. Secondary Outcome: Part 1 and Part 2: Time to Maximum Observed Plasma Concentration (Tmax) of Zanubrutinib
Time Frame: Week 2 Day 1 pre-dose and 24 hours
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 77 | 72
Hours | 2.00 [2.00 to 2.00] | 2.50 [1.08 to 3.00] | 2.00 [1.00 to 3.17] | 2.00 [0.53 to 6.00] | 2.00 [0.33 to 6.00]

9. Secondary Outcome: Part 1 and Part 2: Apparent Terminal Half-life (t1/2) of Zanubrutinib
Time Frame: Week 1 Day 1 pre-dose, 0.5, 1, 2, 3, 4, and 8 hours
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 59 | 18
Hours | 1.94 (28.5) | 1.97 (29.8) | 3.87 (24.9) | 2.73 (60.2) | 3.30 (61.2)

10. Secondary Outcome: Part 1 and Part 2: Apparent Clearance (CL/F) of Zanubrutinib
Time Frame: Week 1 Day 1 pre-dose, 0.5, 1, 2, 3, 4, and 8 hours
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 61 | 18
Liters/hour | 133 (51.5) | 174 (100.6) | 106 (52.7) | 128 (59.4) | 126 (47.8)

11. Secondary Outcome: Part 1 and Part 2: Apparent Volume of Distribution of Zanubrutinib During the Terminal Phase (Vz/F)
Time Frame: Week 1 Day 1 pre-dose, 0.5, 1, 2, 3, 4, and 8 hours
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 61 | 18
Liters | 371 (47.5) | 494 (78.9) | 593 (61.6) | 530 (70.0) | 600 (97.6)

12. Secondary Outcome: Part 1 and Part 2: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with partial or complete response (CR), as assessed by the investigator. For CLL/SLL, ORR includes partial response (PR) with lymphocytosis (PR-L) or better (includes PR-L, PR, nodular PR or nPR and CR with incomplete marrow recovery or CRi) and for MW, ORR includes minor response or better. Efficacy results are reported for each of the B-cell malignancy subtypes: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), Waldenström macroglobulinemia (WM), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), Richter's Transformation (RT), and Hairy cell leukemia (HCL).
Time Frame: Up to 6 years and 7 months
Population: Efficacy Evaluable Set consists of all participants who received at least one dose of zanubrutinib; for WM, participants also must have a baseline IgM (or M-protein) ≥ 5 g/L and no prior exposure to a BTK inhibitor.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part 1 and Part 2: Overall: The dose regimens from Part 1 (40 mg, 80 mg, 160 mg QD, 160 mg BID and 320 mg QD) and Part 2 (160 mg BID and 320 mg QD) were evaluated in different disease types. Efficacy evaluations are reported by disease type for Parts 1 and 2 combined, as pre-specified in the statistical analysis plan.
Arm/Group | Part 1 and Part 2: Overall
Number analyzed (Participants) | 378
Percentage of participants
  CLL/SLL: number analyzed (Participants) | 125
  CLL/SLL | 95.2 [89.8 to 98.2]
  WM: number analyzed (Participants) | 73
  WM | 95.9 [88.5 to 99.1]
  MCL: number analyzed (Participants) | 57
  MCL | 82.5 [70.1 to 91.3]
  MZL: number analyzed (Participants) | 20
  MZL | 85.0 [62.1 to 96.8]
  FL: number analyzed (Participants) | 33
  FL | 36.4 [20.4 to 54.9]
  DLBCL: number analyzed (Participants) | 45
  DLBCL | 42.2 [27.7 to 57.8]
  RT: number analyzed (Participants) | 13
  RT | 61.5 [31.6 to 86.1]
  HCL: number analyzed (Participants) | 12
  HCL | 58.3 [27.7 to 84.8]

13. Secondary Outcome: Part 1 and Part 2: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of participants who achieve a complete response, as assessed by the investigator. For CLL/SLL, CRR includes CRi or better. For WM, CRR includes very good partial response (VGPR) or better. Efficacy results are reported for each of the B-cell malignancy subtypes: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), Waldenström macroglobulinemia (WM), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), Richter's Transformation (RT), and Hairy cell leukemia (HCL).
Time Frame: Up to 6 years and 7 months
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1 and Part 2: Overall
Number analyzed (Participants) | 378
Percentage of participants
  CLL/SLL: number analyzed (Participants) | 125
  CLL/SLL | 16.8 [10.7 to 24.5]
  WM: number analyzed (Participants) | 73
  WM | 46.6 [34.8 to 58.6]
  MCL: number analyzed (Participants) | 57
  MCL | 28.1 [17.0 to 41.5]
  MZL: number analyzed (Participants) | 20
  MZL | 20.0 [5.7 to 43.7]
  FL: number analyzed (Participants) | 33
  FL | 18.2 [7.0 to 35.5]
  DLBCL: number analyzed (Participants) | 45
  DLBCL | 24.4 [12.9 to 39.5]
  RT: number analyzed (Participants) | 13
  RT | 15.4 [1.9 to 45.4]
  HCL: number analyzed (Participants) | 12
  HCL | 16.7 [2.1 to 48.4]

14. Secondary Outcome: Part 1 and Part 2: Partial Response (PR) or Better
Description: PR or better is defined as the percentage of participants who achieve a partial response or better, as assessed by the investigator. For CLL/SLL, includes PR, nPR, CRi, CR and for WM includes PR, VGPR, and CR. Efficacy results are reported for the B-cell malignancy subtypes chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) and Waldenström macroglobulinemia (WM).
Time Frame: Up to 6 years and 7 months
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1 and Part 2: Overall
Number analyzed (Participants) | 385
Percentage of participants
  CLL/SLL: number analyzed (Participants) | 125
  CLL/SLL | 92.0 [85.8 to 96.1]
  WM: number analyzed (Participants) | 73
  WM | 82.2 [71.5 to 90.2]

15. Secondary Outcome: Part 1 and Part 2: Progression-free Survival (PFS)
Description: PFS is defined as the time from the first dose date of study drug to the date of the earliest occurrence of progressive disease or death due to any cause, whichever occurs first. Efficacy results are reported for each of the B-cell malignancy subtypes: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), Waldenström macroglobulinemia (WM), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), Richter's Transformation (RT), and Hairy cell leukemia (HCL).
Time Frame: Up to 6 years and 7 months
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 and Part 2: Overall
Number analyzed (Participants) | 378
Months
  CLL/SLL: number analyzed (Participants) | 125
  CLL/SLL | 61.4 [55.2 to NA] — Data not estimable due to insufficient number of participants with events
  WM: number analyzed (Participants) | 73
  WM | NA [48.9 to NA] — Data not estimable due to insufficient number of participants with events
  MCL: number analyzed (Participants) | 57
  MCL | 27.6 [15.4 to 45.5]
  MZL: number analyzed (Participants) | 20
  MZL | NA [17.1 to NA] — Data not estimable due to insufficient number of participants with events
  FL: number analyzed (Participants) | 33
  FL | 10.4 [7.7 to 22.9]
  DLBCL: number analyzed (Participants) | 45
  DLBCL | 4.1 [2.1 to 5.6]
  RT: number analyzed (Participants) | 13
  RT | 17.3 [2.8 to NA] — Data not estimable due to insufficient number of participants with events
  HCL: number analyzed (Participants) | 12
  HCL | NA [28.7 to NA] — Data not estimable due to insufficient number of participants with events

16. Secondary Outcome: Part 1 and Part 2: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose to death due to any cause. Efficacy results are reported for each of the B-cell malignancy subtypes: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), Waldenström macroglobulinemia (WM), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), Richter's Transformation (RT), and Hairy cell leukemia (HCL).
Time Frame: Up to 6 years and 7 months
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 and Part 2: Overall
Number analyzed (Participants) | 378
Months
  CLL/SLL: number analyzed (Participants) | 125
  CLL/SLL | NA [NA to NA] — Data not estimable due to insufficient number of participants with events
  WM: number analyzed (Participants) | 73
  WM | NA [NA to NA] — Data not estimable due to insufficient number of participants with events
  MCL: number analyzed (Participants) | 57
  MCL | NA [27.2 to NA] — Data not estimable due to insufficient number of participants with events
  MZL: number analyzed (Participants) | 20
  MZL | NA [NA to NA] — Data not estimable due to insufficient number of participants with events
  FL: number analyzed (Participants) | 33
  FL | NA [37.3 to NA] — Data not estimable due to insufficient number of participants with events
  DLBCL: number analyzed (Participants) | 45
  DLBCL | 14.7 [5.5 to 24.8]
  RT: number analyzed (Participants) | 13
  RT | 29.3 [4.2 to NA] — Data not estimable due to insufficient number of participants with events
  HCL: number analyzed (Participants) | 12
  HCL | NA [26.6 to NA] — Data not estimable due to insufficient number of participants with events

17. Secondary Outcome: Part 1 and Part 2: Duration of Response (DOR)
Description: DOR for responders is defined as time from the date of the earliest qualifying response to the date of progressive disease or death for any cause, whichever occurs earlier. Efficacy results are reported for responders (defined as PR or better, except CLL/SLL and WM) in each of the B-cell malignancy subtypes: chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL; PR with lymphocytosis or better), Waldenstrom macroglobulinemia (WM; minor response or better), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), Richter's Transformation (RT), and Hairy cell leukemia (HCL).
Time Frame: Up to 6 years and 7 months
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 and Part 2: Overall
Number analyzed (Participants) | 378
Months
  CLL/SLL: number analyzed (Participants) | 125
  CLL/SLL | 58.6 [52.6 to NA] — Data not estimable due to insufficient number of participants with events
  WM: number analyzed (Participants) | 73
  WM | NA [31.34 to NA] — Data not estimable due to insufficient number of participants with events
  MCL: number analyzed (Participants) | 57
  MCL | 28.2 [16.2 to NA] — Data not estimable due to insufficient number of participants with events
  MZL: number analyzed (Participants) | 20
  MZL | NA [6.5 to NA] — Data not estimable due to insufficient number of participants with events
  FL: number analyzed (Participants) | 33
  FL | NA [8.3 to NA] — Data not estimable due to insufficient number of participants with events
  DLBCL: number analyzed (Participants) | 45
  DLBCL | 14.2 [2.8 to 26.2]
  RT: number analyzed (Participants) | 13
  RT | 25.9 [5.9 to NA] — Data not estimable due to insufficient number of participants with events
  HCL: number analyzed (Participants) | 12
  HCL | NA [NA to NA] — Data not estimable due to insufficient number of participants with events

18. Secondary Outcome: Number of Participants With Greater Than 75% Bruton's Tyrosine Kinase (BTK) Occupancy
Description: Number of participants with greater than 75% BTK occupancy of zanubrutinib in peripheral blood mononuclear cells (PBMCs)
Time Frame: Week 1 Day 1 (W1D1) predose, W1D1 4 hours, W1D2 24 hours, W1D3 predose, and W2D1 predose
Population: Pharmacodynamic analysis set consisted of participants in which PBMCs were collected and evaluable samples were obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
Number analyzed (Participants) | 3 | 4 | 5 | 21 | 10
Participants | 3 | 4 | 5 | 20 | 9

ADVERSE EVENTS:
Time Frame: Up to 6 years and 7 months
Description: One participant in the 320 mg QD group discontinued the study for Other reasons, as shown in the participant flow section, and subsequently died after study discontinuation. That participant is counted under all-cause mortality in this section.
Arm/Group | Part 1: 40 mg QD | Part 1: 80 mg QD | Part 1: 160 mg QD | Part 1 and Part 2: 160 mg BID | Part 1 and Part 2: 320 mg QD
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/4 | 2/5 | 76/278 | 19/95
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/4 | 3/5 | 157/278 | 45/95
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 5/5 | 273/278 | 94/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: 40 mg QD (N=3) | Part 1: 80 mg QD (N=4) | Part 1: 160 mg QD (N=5) | Part 1 and Part 2: 160 mg BID (N=278) | Part 1 and Part 2: 320 mg QD (N=95)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastric volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 9 (12) | 3 (3)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 9 (13) | 3 (5)
Cerebral aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epstein-Barr viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemophilus sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Meningitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (8) | 26 (28) | 6 (6)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scedosporium infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 12 (15) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sarcomatoid carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma of the parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglossal nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic idiopathic pain syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusional disorder, unspecified type (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal artery thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: 40 mg QD (N=3) | Part 1: 80 mg QD (N=4) | Part 1: 160 mg QD (N=5) | Part 1 and Part 2: 160 mg BID (N=278) | Part 1 and Part 2: 320 mg QD (N=95)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 39 (64) | 8 (16)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (3) | 44 (107) | 10 (29)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 25 (42) | 4 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 13 (15) | 3 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 4 (4)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (14) | 3 (3)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Ocular rosacea (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 21 (24) | 8 (11)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (15) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 50 (59) | 23 (29)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (6) | 0 (0) | 77 (122) | 23 (36)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (9) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 24 (27) | 8 (9)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (6) | 1 (1) | 45 (55) | 18 (32)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 4 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (5) | 0 (0) | 29 (38) | 6 (8)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 12 (20) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 49 (55) | 26 (33)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 14 (17) | 11 (11)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 31 (35) | 8 (14)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (13) | 4 (4)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 6 (9)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 36 (85) | 5 (6)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 5 (8)
Cat scratch disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 18 (25) | 11 (15)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 14 (14) | 5 (6)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 3 (7)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 4 (9)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 3 (3)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 13 (15) | 6 (6)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 13 (21) | 9 (10)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 23 (41) | 8 (11)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 22 (32) | 7 (11)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 17 (22) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 22 (24) | 7 (9)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 34 (48) | 8 (14)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 13 (18) | 6 (7)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 2 (7) | 2 (10) | 106 (214) | 46 (89)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 44 (70) | 18 (31)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 3 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 97 (135) | 39 (57)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 28 (38) | 9 (13)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 9 (10)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 5 (7)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 12 (16) | 9 (9)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 4 (8)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 18 (93) | 3 (8)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 17 (28) | 4 (5)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 23 (25) | 6 (6)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 18 (27) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (10) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 37 (54) | 13 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 34 (38) | 23 (28)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 5 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 25 (29) | 12 (13)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 13 (15) | 6 (6)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 17 (19) | 7 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 11 (13) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 5 (5) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 18 (25) | 10 (11)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 22 (45) | 9 (16)
Benign ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 17 (23) | 5 (6)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 28 (35) | 11 (16)
Headache (Nervous system disorders) | 0 (0) | 2 (7) | 2 (2) | 46 (63) | 18 (21)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 13 (14) | 6 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 16 (19) | 4 (6)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (6)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (4)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 18 (19) | 5 (7)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 31 (39) | 12 (15)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 8 (8)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 79 (101) | 21 (24)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 24 (30) | 10 (18)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 27 (44) | 10 (14)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 14 (16) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 19 (27) | 5 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 19 (27) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 5 (6)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (14) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 12 (15) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (13) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 10 (12) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 22 (24) | 9 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 27 (31) | 10 (11)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (10) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 56 (78) | 20 (28)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 9 (12) | 2 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 6 (7)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 15 (17) | 7 (8)
Hypertension (Vascular disorders) | 1 (1) | 1 (3) | 1 (1) | 37 (56) | 11 (15)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT02343120/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02343120/SAP_001.pdf